CLINICAL TRIAL: NCT05552794
Title: Prognostic Value With Combined Sonographic Optic Nerve Sheath Diameter and Near Infrared Spectroscopy Measurements for Predicting Neurological Outcome After Cardiac Arrest
Brief Title: Prognostic Value With Combined ONSD and NIRS Measurements for Predicting Neurological Outcome After Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: Nevsehir Public Hospital (Other Government)
Responsible Party: Principal Investigator, Mehmet Akif Yazar, MD, Assoc. Prof., Nevsehir Public Hospital
Other Study IDs: 2021-1-19
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Cardiac Arrest
Keywords: Cardiac arrest; Optic Nerve Sheath Diameter; Near Infrared Spectroscopy
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Good outcome: Good outcome was defined as cerebral performance category (CPC): 1-2
  Interventions: Diagnostic Test: Optic nerve Sheath Diameter (ONSD)
- Poor outcome: Poor outcome was defined as cerebral performance category (CPC): 3-5
  Interventions: Diagnostic Test: Optic nerve Sheath Diameter (ONSD)

INTERVENTIONS:
Diagnostic Test: Optic nerve Sheath Diameter (ONSD) — ONSD and rSO2 monitoring will perform when the patients arrived in ICU.
  Other Names: Regional cerebral oxygen saturation (rSO2)

SUMMARY:
Cardiac arrest (CA) is a worldwide health problem and is associated with high mortality and morbidity rates. After CA, most patients are exposed to cerebral injury due to anoxic perfusion, resulting in severe neurological deficits. Return of spontaneous circulation (ROSC) after KA causes acute cerebral edema with increased intracranial pressure (ICP) due to ischemia-reperfusion and delayed hyperemia, and deterioration of cerebral perfusion. This reduces the quality of life of most patients after cardiac arrest.

DETAILED DESCRIPTION:
Accurate and early estimation of adverse neurological outcomes in CA survivors is crucial because null treatments for patients who cannot be saved can be avoided. On the contrary, more detailed and comprehensive treatment protocols can be determined for promising patients. In recent years, some studies have focused on the early prediction of neurological outcomes by evaluating the optic nerve sheath diameter (ONSD) of patients after CA. In order to evaluate acute brain edema, ONSD can be measured by computed tomography (CT), and it has been stated in previous studies that changes in gray-white matter ratio (GWR) may be associated with neurological outcomes. However, in addition to CT, ONSD can be easily measured by bedside ultrasonography. Many studies have found a strong association between increased ICP and sonographic ONSD. However, in some studies, it was stated that ONSD measurements were not correlated with neurological outcomes in the 6-month period after ROSC.

On the other hand, Near-Infrared Spectroscopy (NIRS) measures the total oxygen saturation in a given tissue volume by approximating the oxygen saturation of the hemoglobin fraction in the terminal vasculature. With this method, regional oxygen saturation (rSO2) of the brain tissue can be measured noninvasively. In general, post-hypoxic brain injury after cardiac arrest, changes in oxygen consumption, cerebral blood flow or cerebral blood volume may be associated with rSO2 changes in brain tissue. Therefore, using frontal brain rSO2 continuous bedside NIRS monitoring, additional information can be obtained about the early prediction of reliable neurological outcomes. However, some studies show that reliable prognostic results with NIRS monitoring are limited.

Thanks to the combined use of ultrasonography and bedside noninvasive measurements such as ONSD and NIRS, early prediction of the neurological outcomes of cardiac arrest patients with ROSC can positively change the treatment management of this patient group in ICUs with high sensitivity and better neurological outcomes can be achieved.

In this study, the prognostic values of combined ultrasonographic ONSD and NIRS measurements will investigate in predicting neurological outcomes after cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* admitted to the ICU after cardiac arrest,
* GCS ≤6 after arrest,
* age ≥18,
* brain tomography taken within the first 6 hours after the arrest,
* targeted heat management (TTM) applied
* sedated patients

Exclusion Criteria:

* Patients whose measurements could not be made within the first 24 hours after cardiac arrest (early death, major hemodynamic instability, absence of device or investigator at the weekend),
* cardiac arrest due to intracranial trauma or neurological event,
* patients with previous cerebrovascular accident,
* patients who have affected the orbit or eyeball patients with facial trauma,
* patients with ocular pathology such as exophthalmos, glaucoma or cataracts,
* patients who have been or should be sedated,
* those with recurrent CA within three days of ICU admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fourty patients will be enrolled into this investigation.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-12-12 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Cerebral performance category (CPS Scale) | One year
  Cerebral performance category is described as neurological status after cardiac arrest.

SECONDARY OUTCOMES:
Mortality | One year
  After CA,1 year mortality

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Akif Yazar, Principal Investigator — Konya City Hospital
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided